CLINICAL TRIAL: NCT00490269
Title: Phase 1, Pilot Study to Examine the Cardiovascular Effects of Smoked Marijuana, Interactions With Oral Dronabinol, and Effects of Dronabinol on Withdrawal in Marijuana Dependent Volunteers
Brief Title: Ph1 Marinol Interaction Study - Part 2 - 1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, NIDA Project Officer, National Institute on Drug Abuse (NIDA)
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: NIDA-CPU-0013-1
Record Dates: First submitted 2007-06-21; First posted 2007-06-22 (Estimated); Results first posted 2013-04-08 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-08

CONDITIONS: Marijuana Dependence
Keywords: Marijuana dependence
MeSH Terms: conditions — Marijuana Abuse | interventions — Dronabinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Dronabinol (Active Comparator)
  Interventions: Drug: Dronabinol
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo
  Other Names: Placebo comparator arm
  Arms: Placebo
Drug: Dronabinol
  Other Names: Medication intervention
  Arms: Dronabinol

SUMMARY:
This study will examine the effects of oral dronabinol tetrahydrocannabinol (THC) on withdrawal symptoms in marijuana dependent volunteers, and evaluate the safety, pharmacokinetics (PK), and cardiovascular effects of the combination of oral dronabinol and smoked marijuana to determine if there are potential significant drug interactions before conducting outpatient studies.

ELIGIBILITY:
Inclusion Criteria:

* Must be between 18 and 45 years of age
* Must be in good general health and who meet DSM-IV diagnostic criteria for marijuana dependence
* Must be seeking treatment at time of study entry
* Must be able to understand and provide written informed consent
* Must provide 1 marijuana positive urine specimen (> 50 ng/mL) within the 28-day screening period
* If female and of child bearing potential, agrees to use birth control.

Exclusion

Criteria:

* Please contact site for more information

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2006-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Louis Cantilena, M.D., Principal Investigator — Uniformed Services University of Health Science
Locations (1):
- Uniformed Services University of Health Science, Bethesda, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was from October 31, 2006 to December 5, 2007. The study was conducted at the NIDA funded clinical pharmacology unit (CPU) at Uniformed Services University for the Health Sciences (USUHS).
Pre-assignment Details: Volunteers meeting the maximum 28-day screening assessment period and eligibility criteria were enrolled into the Phase-1 clinical trial. The subjects had to meet the following criteria to be eligible: be non-treatment seeking, experienced marijuana users with dependence for the past year, and subjects that were in good general health.
Groups:
- Dronabinol; Placebo: Subjects received either 10mg of study drug or matched placebo capsules 5 times per day on non-smoking Days 4-8 at approximately 0800, 1100, 1400, 1700 and 2000 hours. On day 9, study drug (or placebo)was given only 3 times at the 1100 and 1400 hour time points. On day 10, only the first dose of study drug (or placebo) was given at 0800.
Period: Dronabinol Then Placebo
Arm/Group | Dronabinol | Placebo
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Placebo Then Dronabinol
Arm/Group | Dronabinol | Placebo
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dronabinol | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 12
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.2 (3.6) | 27.2 (4.9) | 27.2 (4.3)
Gender [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Experience Cardiovascular Effects of Smoked Marijuana or Has Any Other Combination Side Effects.
Description: Does dronabinol (when given during smoking of a marijuana cigarette) show changes in the number of participants that experience cardiovascular effects of smoked marijuana or has any other combination side effects.
Time Frame: Day 9 and 10
Measure: Number; unit: participants
Arm/Group | Dronabinol | Placebo
Number analyzed (Participants) | 6 | 6
participants | 6 | 6

ADVERSE EVENTS:
Time Frame: Adverse events were collected starting on Day 0 through Day 12
Description: If a subject experienced more than one adverse events (AE), it would be recorded as a separate AE.
Arm/Group | Dronabinol | Placebo
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/6
Other Adverse Events (participants affected / at risk) | 6/6 | 1/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dronabinol (N=6) | Placebo (N=6)
Anxiety Disorder (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dronabinol (N=6) | Placebo (N=6)
Palpitations (Cardiac disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 — Mild adverse event; possibly related to study drug.
Fatigue (General disorders) | 1 | 0 — Mild adverse event; possibly related to study drug.
Catheter site hemmorage (General disorders) | 1 | 0
Catheter site adema (General disorders) | 1 | 0
Injection site inflammation (General disorders) | 1 | 0
Transamenase Increase (Hepatobiliary disorders) | 1 | 0 — Moderate adverse event; possibly related to study drug.
Decrease in Appetite (NOS) (Metabolism and nutrition disorders) | 1 | 0 — Mild adverse event; possibly related to study drug.
Headache (Nervous system disorders) | 1 | 0 — Mild adverse event; possibly related to study drug.
Syncope (Nervous system disorders) | 1 | 0 — Moderate adverse event, remotely related to study drug.
Insomnolence (Nervous system disorders) | 1 | 0 — Mild adverse event; possibly related to study drug.
Anxiety (Psychiatric disorders) | 1 | 0 — Moderate adverse even; probably related to study drug.
Anxiety disorders and symptoms (Psychiatric disorders) | 1 | 0 — Mild adverse event; possibly related to study drug.
Irritability (Psychiatric disorders) | 1 | 0 — Mild adverse event; possibly related to study drug.
Polymenorrhea (Reproductive system and breast disorders) | 1 | 0 — Mild adverse event and possibly related to study drug.
Lip ulceration (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No